CLINICAL TRIAL: NCT05182905
Title: A Phase 0/1b, Single Center, Clinical Trial With an Expansion Phase of AZD1390 Plus Fractionated Radiotherapy in Recurrent and Newly Diagnosed WHO Grade 4 Glioma Patients
Brief Title: AZD1390 in Recurrent and Newly Diagnosed WHO Grade 4 Glioma Patients
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nader Sanai (Other)
Collaborators: Barrow Neurological Institute (Other); Ivy Brain Tumor Center (Other); AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Nader Sanai, Director of the Ivy Brain Tumor Center, St. Joseph's Hospital and Medical Center, Phoenix
Organization: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ivy 2020-10
Record Dates: First submitted 2021-12-22; First posted 2022-01-10 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Glioblastoma; Glioma; Glioblastoma Multiforme; Glioma, Malignant
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — AZD1390

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A: Recurrent Grade 4 Glioma Surgical Cohort Time Escalation (Experimental)
  Interventions: Drug: AZD1390
- Arm B: Recurrent Grade 4 Glioma Dose Escalation (Experimental)
  Interventions: Drug: AZD1390
- Arm C: Newly-diagnosed Grade 4 Glioma (Experimental)
  Interventions: Drug: AZD1390

INTERVENTIONS:
Drug: AZD1390 — Phase 0: AZD1390 administered orally daily for 3 days prior to resection
  Phase 1b: AZD1390 administered daily for 5 days concurrently with standard of care radiation therapy

SUMMARY:
This is an open-label, single-center Phase 0/1b study that will enroll at least 27 participants with recurrent WHO Grade 4 Glioma requiring re-radiation and approximately 35 participants with newly-diagnosed WHO Grade 4 glioma (nGBM). The trial will be composed of a Phase 0 component (subdivided into Arms A - C), and an expansion Phase 1b. Patients with tumors demonstrating a positive PK response in the Phase 0 component of the study will be eligible to graduate to an expansion phase that combines therapeutic dosing of AZD1390 plus standard-of-care fractionated radiotherapy (RT).

ELIGIBILITY:
Inclusion Criteria:

1a. Arm C only: Participants undergoing resection for a suspected newly diagnosed WHO Grade 4 glioma. Participants will also need to have radiation planned as part of the post-surgical treatment plan; OR,

1b. Arms A and B only: Participants who have had a prior resection of diagnosed glioma (2021 WHO grade IV), defined as participants who have progressed on or following standard therapy, which includes maximal surgical resection, temozolomide, and fractionated radiotherapy. Participants will also need to have radiation planned as part of the post-surgical treatment plan.

2. Participants must have measurable disease preoperatively, defined as at least 1 contrast-enhancing lesion, with 2 perpendicular measurements of at least 1 cm.

3. Provision of signed and dated, written informed consent (personally or by the legally authorized representative, if applicable) prior to any study specific procedures, sampling and analyses.

4. Age ≥18 at time of consent. 5. Have a performance status (PS) of ≤2 on the Eastern Cooperative Oncology (Group (ECOG) scale1.

6. Ability to swallow oral medications. 7. Participant has adequate bone marrow and organ function as defined by the following laboratory values (as assessed by the local laboratory for eligibility):

* Adequate bone marrow function:

  * absolute neutrophil count ≥1,500/mcL
  * Platelets (at time of surgery) ≥100,000/mcL
  * hemoglobin ≥9.0 g/dL Participants may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin earlier than the day after the erythrocyte transfusion.
* Adequate hepatic function:

  o total bilirubin ≤1.5 X ULN. Participants with Gilbert's syndrome with a total bilirubin ≤2.0 times ULN and direct bilirubin within normal limits are permitted.

  o AST(SGOT) ≤2.5 X institutional ULN

  o ALT(SGPT) ≤2.5 X institutional ULN
* Adequate pancreatic function:

  o Amylase within normal limits (WNL)

  o Lipase within normal limits (WNL)
* Adequate renal function:

  * Serum creatinine ≤1.5 X ULN or estimated creatinine clearance ≥ 60 mL/min (calculated using Institutional standard method) 8. Participants with tumor-induced seizures must be well-controlled on a stable anti-epileptic treatment.

    9. Participants must be willing to receive prophylaxis with levetiracetam for the duration of study drug administration (or alternative anti-epileptic if agreed with Medical Monitor) 10. Confirmed negative serum pregnancy test (β-hCG) before starting study treatment or participant who is no longer of childbearing potential due to surgical, chemical, or natural menopause.

    11. For females of reproductive potential: use of highly effective contraception and agreement to use such a method during study participation until the end of treatment administration and for 16 weeks after the last dose of study drug.

    12. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner until the end of treatment administration and for 16 weeks after the last dose of study drug.

    13. Agreement to adhere to Lifestyle Considerations (see Section 5.3) throughout study duration.

Exclusion Criteria:

1. Current use of coumarin-derived anticoagulant for treatment, prophylaxis or otherwise, that cannot be discontinued prior to surgery. Therapy with heparin, low molecular weight heparin (LMWH) or fondaparinux is allowed.
2. Pregnancy or lactation.
3. Known allergic reactions to components of the AZD1390.
4. Known to have active (acute or chronic) or uncontrolled severe infection, liver disease such as cirrhosis, decompensated liver disease, and active and chronic hepatitis, as determined by the investigator.
5. Known active systemic bacterial infection (requiring intravenous [IV] antibiotics or fever >38.5°C at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]. Screening of viral infection is not required for enrollment.
6. The participant has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.
7. Any of the following cardiac criteria:

   * Cardiac dysfunction defined as: Myocardial infarction within six months of study entry, NYHA Class II/III/IV heart failure, unstable angina or unstable cardiac arrhythmias.
   * Mean resting corrected QT interval (QTcF) > 470 msec obtained from 3 electrocardiograms (ECGs) (QTc interval will be calculated using Fridericia's formula).
   * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG, e.g., complete left bundle branch block, third degree heart block.
   * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years-of-age. Patients stable on concomitant medications known to prolong the QT interval may be allowed to participate in the study provided that their mean resting corrected QT interval (QTcF) is < 470 msec at baseline and after discussion with the Medical Monitor.
8. History of epileptic disorder or any seizure history unrelated to tumor.
9. History or presence of myopathy or raised creatine kinase (CK) >5 x upper limit of normal (ULN) on 2 occasions at screening.
10. Past medical history of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
11. Participant has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
12. Prior therapy with ATM kinase inhibitors.
13. Treatment with strong inhibitors or inducers of CYP3A4 within 2 weeks prior to receiving study drug.
14. Prior treatment with pneumotoxic drugs, e.g. busulfan, bleomycin, within the past year. If prior therapy in lifetime, then excluded if history of pulmonary toxicities from administration. Patients who have received treatment with nitrosoureas (e.g., BCNU, CCNU) in the year before study entry without experiencing lung toxicity are allowed on study.
15. Treatment with another investigational drug or other intervention within 5 half-lives of the investigational product, whichever is longer.
16. With the exception of alopecia, any unresolved toxicities from prior therapy greater than National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v5.0) Grade 1 at the time of starting study treatment and patients with chronic Grade 2 unresolved toxicities may be eligible following discussion with the Medical Monitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2022-03-09 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Phase 0: The relative pharmacokinetics (PK) of AZD1390 in tumor tissue from Grade 4 glioma participants treated with AZD1390 | Phase 0 Intraoperative
  For PK analysis, total and unbound AZD1390 concentration in Gd-enhancing and Gd-non-enhancing tumor tissue.
Phase 1b: Examine the rate of 6-month progression-free survival glioma participants with demonstrated PK effect. | From the date of Phase 0 surgery to the date of progression
  The rate of 6-month progression-free survival (PFS6) measured from time of surgery to date of recurrence or death, whichever occurs first, will be summarized.

SECONDARY OUTCOMES:
Phase 0: To evaluate the relative pharmacokinetics (PK) of AZD1390 in CSF | Phase 0 Intraoperative
  AZD1390 level in CSF will be determined.
Drug-related toxicity | Through study completion, an average of once a week
  Incidence of drug-related toxicity
Adverse events | Through study completion, an average of once a week
  Number of adverse events through study completion
Deaths | Every 3 months for up to 12 months after completing study treatment
  Number and incidence of deaths
Incidence of clinical laboratory abnormalities per CTCAE | Through study completion, an average of once a week
  Number of clinical laboratory abnormalities per CTCAE
Phase 1b: Overall survival | From the date of Phase 0 surgery to the date of death due to any cause
  Median overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Nader Sanai, MD, Principal Investigator — Chief Scientific Officer/Director
Locations (1):
- St. Joseph's Hospital and Medical Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Ivy Brain Tumor Center Website — http://ivybraintumorcenter.org